CLINICAL TRIAL: NCT05680974
Title: Gewinnung, Kultur Und Studien Von primären Humanen Zelltypen, Geweben Und Blut für Die Gezielte Behandlung Von Seltenen Hauterkrankungen
Brief Title: Personalized Therapy of Patients Suffering From Rare Genodermatoses
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Principal Investigator, Wolfram Hoetzenecker, Chair of the Department of Dermatology and Venerology, Johannes Kepler University of Linz
Other Study IDs: RAREDISEASE
Record Dates: First submitted 2023-01-02; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Rare Diseases
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and skin biopsy samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: If a targetable cytokine is increased in the lesional skin of a patient, this patient is treated with the respective antibody therapy (off-label use of approved drug). — If a targetable cytokine is increased in the lesional skin of a patient, this patient is treated with the respective antibody therapy (off-label use of approved drug).

SUMMARY:
Rare skin diseases are generally defined as serious life-threatening, progressive chronic diseases of the skin that occur extremely rarely (i.e., 5 in 10,000 people are affected). More than 80% are hereditary. In most cases, late diagnosis and the lack of therapeutic strategies also contribute to severe disease progression. Therefore, new therapeutic options are urgently needed and with them knowledge of the underlying mechanisms of disease development.

The aim of this project is to better understand disease mechanisms and to identify new pathways and drug targets that will improve patient care or therapy. In order to investigate the mechanisms of disease development, it is necessary to isolate biological material, i.e. blood and affected skin tissue from patients. For this purpose, adults 18 years of age and older with a congenital rare skin disease are included. We take blood and (lesional) skin biopsies from patients to perform immunoprofiling, as well as cell biological studies with the patient's cells. The risk for the patients is low, as only peripheral blood and skin biopsies are taken. Potential risks include bruising and pain as well as infection, postoperative bleeding, wound infection or delayed wound healing, pain, and scarring.

The samples are pseudonymized and stored with the pseudonym only. Cells and skin samples are only preserved with the prior consent of the patient.

ELIGIBILITY:
Inclusion Criteria:

* age of 18
* rare disease is known or suspected
* patent consent

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from rare genodermatoses.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of disease as assessed by affected body surface area by 50 % upon off-label treatment with approved monoclonal antibody therapies | 12 months
  Severely affected consenting patients will be treated with approved monoclonal antibodies targeting exactly the cytokines that are increased in the patient's lesional skin.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Ettinger, MD PhD, Study Chair — Kepler University Hospital Linz
Locations (1):
- Kepler University Hospital Linz, Linz, Austria

IPD SHARING:
Plan to Share IPD: Undecided